CLINICAL TRIAL: NCT06312826
Title: A Prospective Randomized Comparative Cohort Study to Investigate Abbreviated Magnetic Resonance Imaging Using Gadoxetic Acid and Ultrasonography for Surveillance of Early-stage HCC in Patients at High Risk for HCC
Brief Title: Abbreviated MRI Using Gadoxetic Acid Versus Ultrasonography for Surveillance of Early-stage HCC in Patients at High Risk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, So Yeon Kim, MD, PhD, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KCT0007417; 2022-0661 (Other: Asan Medical Center Institutional Review Board)
Record Dates: First submitted 2024-03-09; First posted 2024-03-15 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Liver Cirrhosis; Hepatocellular Carcinoma
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US group (Active Comparator): Subjects will be evaluated by two rounds of tests with abdominal US for the surveillance of HCC at intervals of 6 months.
  Interventions: Procedure: Abdominal US
- AMRI group (Experimental): Subjects will be evaluated by two rounds of tests with AMRI for the surveillance of HCC at intervals of 6 months.
  Interventions: Procedure: AMRI

INTERVENTIONS:
Procedure: Abdominal US — The acquired images included B-mode images of the left hepatic lobe through transverse and longitudinal scans including images of the umbilical portion of the left portal vein, and images of the right hepatic lobe through subcostal and intercostal scans including images of the right hepatic dome, right portal vein, and right hepatic vein with additional images of the confluence of both portal vein and three hepatic veins. When a liver observation was seen, additional images were taken, and its diameter was measured on both transverse and longitudinal planes.
  Arms: US group
Procedure: AMRI — The study subjects receive intravenous injection of gadoxetic acid (0.025 mmol/kg, Primovist; Bayer, Berlin, Germany) in the waiting room and then proceed to the examination room for MRI testing 15-20 minutes later. The MRI examination is conducted using a 3T MRI machine, and the MRI protocol consists of T2-weighted imaging, diffusion-weighted imaging (b value of 0, 50, and 500 s/mm2), and hepatobiliary phase imaging.
  Arms: AMRI group

SUMMARY:
Hepatocellular carcinoma (HCC) is the third most frequent cause of cancer-related deaths worldwide. The incidence of HCC has been rapidly rising worldwide over the last two decades. In order to improve survival with curative treatment, regular surveillance to detect early-stage HCC is recommended for at-risk populations. Although ultrasonography (US) has been endorsed as the primary surveillance tool for HCC, a recent meta-analysis found that US has a sensitivity of 47% for detecting early-stage HCC, and its sensitivity for detecting early-stage HCC has been questioned. Many recent studies have explored the potential of alternative surveillance tools for HCC other than US, particularly for high-risk patients. Although complete gadoxetic acid-enhanced magnetic resonance imaging (MRI) demonstrated excellent performance, its high cost and long examination time can hamper its widespread adoption. Abbreviated MRI (AMRI) including hepatobiliary-phase imaging is a promising option to detect potential indicators of HCC, maintaining the benefits of highly sensitive imaging while reducing the examination time by omitting dynamic contrast-enhanced imaging. Because US is the current primary surveillance tool for HCC, this new surveillance tool must be compared with US in a prospective randomized comparative design.

Thus, the hypothesis to be proved in this study is as follows: AMRI with gadoxetic acid will show a significantly higher detection rate compared to US for the detection of early-stage HCC in patients with cirrhosis and at high risk of developing HCC, defined as an estimated annual HCC risk of higher than 5%. We will also analyze whether the false-referral rate of AMRI with gadoxetic acid is not compromised by its high detection rate.

DETAILED DESCRIPTION:
A total of 806 subjects will be randomized in a 1:1 ratio into the US group and the AMRI group. Subjects will be evaluated by two rounds of tests with US or AMRI at intervals of 6 months. After the completion of the two evaluation rounds, at least 6 months of clinical follow-up data will be collected to record the occurrence of interval cancer.

US group: Subjects will be evaluated by two rounds of tests with abdominal US for the surveillance of HCC at intervals of 6 months.

AMRI group: Subjects will be evaluated by two rounds of tests with AMRI with gadoxetic acid for the surveillance of HCC at intervals of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with liver cirrhosis who are classified as high-risk for HCC "High-risk for HCC" is defined as exceeding 2.33 according to the following formula, taking into consideration previous research results: Risk Index = 1.65 (if the prothrombin activity is ≤75%) + 1.41 (if the age is 50 years or older) + 0.92 (if the platelet count is <100 x 10^3/mm^3) + 0.74 (if the presence of anti-HCV or HBsAg is positive)

   Liver cirrhosis is diagnosed when it occurs within the 12 months prior to the research examination, regardless of the cause. The diagnostic criteria for liver cirrhosis are as follows:

   Diagnosis of liver cirrhosis histologically by liver tissue examination, Showing a value of 12 kPa or higher in liver stiffness measurement (fibroscan), Showing typical features of liver cirrhosis on imaging examination or evidence of portal hypertension such as splenomegaly or varices on imaging examination.
2. Absence of previous or current history o f HCC within 6 months prior to screening
3. Eastern Cooperative Oncology Group performance status of 0-2
4. Patient is able to comply with scheduled visits, evaluation plans, and other study procedures
5. Patient is willing to provide written informed consent

Exclusion Criteria:

1. Active or suspected cancer, or a history of malignancy where the risk of recurrence is equal or higher than 20% within 2 years.
2. Significant medical comorbidities in which survival is predicted to be less than 3 years
3. Estimated glomerular filtration rate < 30 mL/min/1.73m²
4. Patient not eligible for applying LI-RADS criteria, such as Budd-Chiari Syndrome
5. Precautions for MRI (cardiac pacemaker, severe claustrophobia that may interfere with protocol compliance).
6. Any other condition which, in the opinion of the Investigator, would make the patient unsuitable for enrollment or could interfere with completing the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Estimated)
Dates: Start 2022-08-26 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate of patients with early stage HCC | 6 months after the completion of the 2 surveillance rounds
  Detection rate = TP / TP + FP +TN + FN

SECONDARY OUTCOMES:
False referral rate of patients with early stage HCC | 6 months after the completion of the 2 surveillance rounds
  False referral rate = FP / TP +FP +TN + FN
Detection rate of patients with very early stage HCC | 6 months after the completion of the 2 surveillance rounds
  Detection rate = TP / TP + FP +TN + FN
False referral rate of patients with very early stage HCC | 6 months after the completion of the 2 surveillance rounds
  False referral rate = FP / TP +FP +TN + FN
Detection rate of patients with all-stage HCC | 6 months after the completion of the 2 surveillance rounds
  Detection rate = TP / TP + FP +TN + FN
False referral rate of patients with all-stage HCC | 6 months after the completion of the 2 surveillance rounds
  False referral rate = FP / TP +FP +TN + FN
Stage distribution at initial HCC diagnosis | At the time of diagnosis
  Distribution of BCLC stage (0, A, B, and C)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park HJ, Choi J, Kim DW, Choi SH, Choi WM, Chung SW, Lee D, Shim JH, Lee HC, Lim YS, Kim MJ, Singal AG, Park SH, Kim SY. Abbreviated gadoxetic acid-enhanced MRI versus ultrasonography for HCC surveillance in high-risk patients: A randomized trial protocol. Hepatol Commun. 2025 Dec 1;9(12):e0839. doi: 10.1097/HC9.0000000000000839. eCollection 2025 Dec 1. PMID 41481895